CLINICAL TRIAL: NCT00587054
Title: Phase II Trial of Allogeneic T-Cell Depleted Hematopoietic Stem Cell Transplants From HLA Compatible, Related and Unrelated Donors After a Myeloablative Preparative Regimen With Hyperfractionated TBI, Thiotepa and Fludarabine For Treatment of Adult Patients (>18 Years) With Lymphohematopoietic Disorders
Brief Title: Trial of Allogeneic Stem Cell Transplants From HLA Compatible, Related and Unrelated Donors After a Myeloablative Preparative Regimen With Hyperfractionated TBI, Thiotepa and Fludarabine For Adult Patients With Lymphohematopoietic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-070; CA23766; CA33049
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Allogeneic Stem Cell Transplant; Leukemia; Non-Hodgkins; Lymphoblastic Lymphoma; Myelodysplastic Syndrome; Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: leukemia; non-Hodgkins; lymphoblastic lymphoma; myelodysplastic syndrome; paroxysmal nocturnal hemoglobinuria (PNH); cytoreductive regimen; allogeneic stem cell transplant
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Hemoglobinuria, Paroxysmal

ARMS (1):
- Transplant Patients (Experimental)
  Interventions: Drug: cytoreductive regimen followed by a CD34+E- selected allogeneic stem cell transplant

INTERVENTIONS:
Drug: cytoreductive regimen followed by a CD34+E- selected allogeneic stem cell transplant — Myeloablative and will consist of hyperfractionated TBI - 1375 cGy administered in 11 doses of 125 cGy each over a total of four days, with three doses on three days and two doses on the last day, fludarabine 25 mg/m2 IV x 5 days, and thiotepa 5mg/kg IV x 2 days. Recipients of HLA identical related transplants will not receive ATG to promote engraftment. Recipients of HLA mismatched related or unrelated stem cells will receive ATG for two days prior to the transplant. G-CSF mobilized CD34+E- PBSCs obtained from the HLA compatible donor will be infused on day 0. Post transplantation G-CSF will be administered only if clinically indicated and should begin on or after d+7.
  Patients will be clinically evaluated at each clinic visit for incidence and severity of acute and chronic GVHD and transplant associated morbidity. Sequential evaluation of functional reconstitution of hematopoiesis and immunity will be made as per the BMT Service guidelines.

SUMMARY:
This is a phase II, single-center study to evaluate the efficacy of a novel cytoreductive regimen followed by CD34+E- selected T cell depleted allogeneic stem cell (or soybean agglutinated and E-rosetted BM) transplant as treatment for patients with acute and chronic leukemias, lymphoma and myelodysplstic syndrome/PNH. The impact of the change in conditioning regimen and use of CD34-selected T cell depleted PBSCs on transplanted related morbidity and mortality and disease free survival will be assessed.

DETAILED DESCRIPTION:
The purpose of this study is: (1) to try to kill any cancer or precancer cells that are in your body, and to reduce the side effects of a transplant, which we have seen in our previous studies, (2) to see if this treatment with a new recipe of radiation and chemotherapy can suppress your immune system enough for the stem cells to 'take' and grow, (3) to see if the specially prepared stem cells can grow in you without a problem called graft-versus-host disease (GvHD) occurring.

One of the major side effects of any stem cell transplant is a condition known as graft vs. host disease or GVHD. GVHD is an immune reaction caused by certain cells from the transplanted stem cells called T-lymphocytes (or T-cells). The T-cells from your donor may see your organs as foreign and attack them. New ways to remove the T-cells from the stem cells before the transplant are being used to try and prevent GVHD. In some studies, the removal of T-cells from the stem cells has been successful for many patients in preventing both short-term (acute) and long-term (chronic) forms of GVHD. However, the removal of T-cells may increase the chance that the new bone marrow developing from the stem cells will be rejected or will not function well. Rejection of the transplant means that some of your own cells have survived the chemo and radiation therapy, and are attacking the new bone marrow cells. This condition can be lifethreatening because of an increased risk of infections and bleeding and would require your getting more treatment and additional stem cells. Studies like this one are designed to find better ways to avoid GVHD without increasing the risk of other problems such as graft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven acute or chronic leukemia, non Hodgkins and lymphoblastic lymphoma or myelodysplastic syndrome
* HLA 6/6 or 5/6 antigen matched related or unrelated donor
* creatinine = normal or if not, CrCl > 60 ml/min/1.73ml
* total bilirubin < 2.5, AST < 2xnl, cardiac function > 50%
* pulmonary function - asymptomatic or if not DLCO > %50% (corrected for Hgb)
* Karnofsky performance status > 70%
* negative pregnancy test (where applicable)
* signed informed consent of patient and donor.

Exclusion Criteria:

* Pregnancy or lactation
* unwillingness to comply with protocol treatment or follow-up
* uncontrolled infection
* HIV or HTLV positivity
* active CNS/skin disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2001-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Jakubowski, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant Patients: Adult Patients (>18 years) with Lymphohematopoietic Disorders will receive Allogeneic T-Cell Depleted Hematopoietic Stem Cell Transplants After a Myeloablative Preparative Regimen With Hyperfractionated TBI, Thiotepa and Fludarabine
Period: Overall Study
Arm/Group | Transplant Patients
Started | 129
Completed | 120
Not Completed | 9
Not completed — Patient not treated | 9

BASELINE CHARACTERISTICS:
Arm/Group | Transplant Patients
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 127
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Transplant Patients
Description: Calculate the median overall survival of transplant patients
Time Frame: up to 6 years
Measure: Median (Full Range); unit: Days
Arm/Group | Transplant Patients
Number analyzed (Participants) | 120
Days | 727.5 [12 to 2231]

ADVERSE EVENTS:
Arm/Group | Transplant Patients
Serious Adverse Events (participants affected / at risk) | 13/129
Other Adverse Events (participants affected / at risk) | 126/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Patients (N=129)
Adult respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Constitutional symptoms, other (General disorders) | 4 (4)
Hemorrhage, other (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Musculoskeletal and connective tissue disorders) | 3 (3)
infection unknown absolut neutriphil counts (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 3 (3)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Vision-double vision (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Patients (N=129)
Alkaline phosphatase (Metabolism and nutrition disorders) | 23 (23)
Bilirubin (Metabolism and nutrition disorders) | 31 (31)
Creatinine (Metabolism and nutrition disorders) | 13 (13)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 117 (117)
Hyperglycemia (Metabolism and nutrition disorders) | 58 (58)
Hyperkalemia (Metabolism and nutrition disorders) | 26 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 35 (35)
Hypokalemia (Metabolism and nutrition disorders) | 60 (60)
Hyponatremia (Metabolism and nutrition disorders) | 35 (35)
Hypophosphatemia (Metabolism and nutrition disorders) | 48 (48)
Leukocytes (Blood and lymphatic system disorders) | 125 (125)
Lymphopenia (Blood and lymphatic system disorders) | 125 (125)
Neutrophils (Blood and lymphatic system disorders) | 123 (123)
Platelets (Blood and lymphatic system disorders) | 124 (124)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 11 (11)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 22 (22)
SGOT (AST) (Blood and lymphatic system disorders) | 28 (28)
SGPT (ALT) (Blood and lymphatic system disorders) | 42 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No